CLINICAL TRIAL: NCT06117852
Title: Chronic Kidney Disease Registry Platform Study
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00355
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants with CKD and High Proteinuria
- Group B: Participants with CKD and Hypertension

SUMMARY:
This is a multicenter, prospective, observational registry platform study which is designed to establish a CKD registry platform by collecting data on the demographics, etiology and staging, clinical characteristics, diagnostic and treatment patterns, and clinical outcomes of patients with chronic kidney disease (CKD), to describe the current status of the diagnosis and treatment of patients with CKD and the gaps from the diagnostic and treatment guidelines, explore the risk factors for disease progression and clinical outcomes in CKD patients, and construct a risk prediction model for CKD progression and clinical outcomes

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is characterized by its high prevalence, low awareness, poor prognosis, and high medical costs, which seriously jeopardize human health. High-risk factors such as severe proteinuria and uncontrolled hypertension further exacerbate the progression of CKD, leading to adverse kidney outcomes, cardiovascular diseases, hospitalizations, and increased mortality. Given these challenges, establishing a registry platform for high-risk CKD patients in China is essential.

This multicenter, prospective, observational registry study aims to comprehensively gather data on the demographic and clinical characteristics, diagnosis and treatment patterns, clinical outcomes, and healthcare resource utilization among high-risk CKD patients in China, which will facilitate the exploration of risk factors associated with CKD progression and clinical outcomes and support the development of predictive models for these outcomes. During the study period from 2023 to 2027, we plan to enroll approximately 5,000 Chinese CKD patients across at least 37 study sites. The study will establish different CKD subpopulations, including but not limited to CKD with High Proteinuria and CKD with Hypertension. Baseline data and annual follow-up data will be collected for the enrolled CKD patients. By establishing this CKD registry platform, we aim to describe the current status of the diagnosis and treatment of CKD patients, identify gaps from diagnostic and treatment guidelines, explore risk factors for disease progression and clinical outcomes, and construct risk prediction models for CKD progression and clinical outcomes.

ELIGIBILITY:
Registry Platform Study Basic Inclusion & Exclusion Criteria:

Inclusion Criteria:

1. Aged ≥ 18 years at enrollment;
2. Patients who meet the diagnostic criteria for CKD;
3. Last eGFR ≥ 20 and < 90 mL/min/1.73 m2 (with the CKD-EPI formula) within 12 months prior to enrollment;
4. Patients who voluntarily participate in this study and has signed and dated the informed consent form for the study;

Exclusion Criteria:

1. Patients who have previously undergone/are undergoing/are planning to undergo solid organ transplantation;
2. Patients with active malignant tumor requiring drug therapy at the time of screening;
3. Women who are pregnant, planning to become pregnant or who are breastfeeding.

Group A (Participants with CKD and High Proteinuria) Inclusion & Exclusion Criteria:

Inclusion criteria:

Last documented proteinuria test within 12 months prior to enrollment indicating UACR ≥ 700 mg/g, or UPCR ≥ 1000 mg/g, or 24 h urine protein (quantitative) ≥ 1 g/24 h.

Exclusion criteria:

1. Patients with NYHA class III or IV heart failure at screening;
2. Patients who have had myocardial infarction, unstable angina, stroke, transient ischemic attack (TIA), or undergone cardiac surgery, percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), valvular repair/replacement, or received treatment with left ventricular assist device within 3 months prior to screening;
3. Patients undergoing renal replacement therapy (RRT) at screening;
4. Patients on systemic immunosuppression at screening (inhalation, intranasal administration, or topical steroids are allowed) except for stable maintenance therapy. The stable maintenance therapy means treatment at least 3 months with Prednisone 10mg/day or lower (or equivalent dose of other drugs), Azathioprine 100mg/day or lower, or Mycophenolate mofetil 1000mg/day or lower (or equivalent dose of other drugs);
5. Patients with a life expectancy of less than 1 year, as judged by the investigator;
6. Patients who have participated in another interventional clinical trial and have received the investigational drug within 1 month prior to being enrolled.

Group B (patients with CKD and Hypertension) Inclusion & Exclusion Criteria:

Inclusion criteria:

1. Last documented test within 12 months prior to enrollment indicating UACR>200 mg/g（22.6 mg/mmol）and <5000 mg/g（565 mg/mmol）, or UPCR >500 mg/g and <8000 mg/g, or 24 h urine protein (quantitative) >0.5 g/24 h and <8 g/24 h;
2. Patients with hypertension history and Systolic Blood Pressure ≥130 mmHg at screening;

Exclusion criteria:

1. Patients with NYHA class IV heart failure at screening;
2. Patients who have had stroke, transient ischemic attack (TIA), Carotid artery surgery or carotid angioplasty and stenting, acute Coronary Syndrome, or hospitalization caused by heart failure deterioration within 3 months prior to screening;
3. Patients who have known severe hepatic injury (defined as Child-Pugh class C) based on medical history;
4. Patients undergoing renal replacement therapy (RRT) within 12 weeks prior to screening;
5. Patients on systemic immunosuppression prior to screening (inhalation, intranasal administration, or topical steroids are allowed) except for stable maintenance therapy at least 3 months;
6. Patients with a life expectancy of less than 1 year, as judged by the investigator;
7. Patients who have participated in another interventional clinical trial and have received the investigational drug within 1 months prior to being enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD patients with age not less than 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease Progression in CKD Patients | From 2023 to 2027
  Patients with progressive deterioration of renal function, including decreased eGFR, rapid progression of CKD
Clinical Outcomes in CKD Patients - Renal Outcomes | From 2023 to 2027
  Including renal transplantation, maintenance dialysis, death from renal failure, persistent low eGFR, persistent percent decline in eGFR
Clinical Outcomes in CKD Patients - Cardiovascular Outcomes | From 2023 to 2027
  Including acute myocardial infarction, sudden serious arrhythmia, hospitalization due to heart failure, stroke or apoplexy, cardiovascular death
Clinical Outcomes in CKD Patients - Cardiac and Renal Composite Outcomes | From 2023 to 2027
  Composite outcome measure consisting of multiple single outcome measures for cardiovascular outcomes and renal outcomes
Clinical Outcomes in CKD Patients - All-cause Mortality | From 2023 to 2027
  In-hospital or out-of-hospital deaths from all causes, including but not limited to deaths related to cardiovascular outcomes or renal outcomes, etc.
Changes in Patient Conditions - Changes in Proteinuria | From 2023 to 2027
  Changes in UACR, UPCR, and 24 h urine protein (quantitative) from baseline
Estimates of Changes in Patient Conditions - Changes in eGFR | From 2023 to 2027
  Changes from baseline in glomerular filtration rate (eGFR), eGFR slope

CONTACTS AND LOCATIONS:
Overall Officials: Bicheng Liu, Principal Investigator — Zhongda Hospital
Locations (34):
- China (34):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Huaian
  - Research Site, Jilin
  - Research Site, Jining
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Panjin
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenzhen
  - Research Site, Taizhou
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xiamen
  - Research Site, Xianyang
  - Research Site, Yantai
  - Research Site, Yibin
  - Research Site, Zhongshan
  - Research Site, Zhuzhou
  - Research Site, Zigong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Access Criteria: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.